CLINICAL TRIAL: NCT03545113
Title: A Randomized Pilot Study Comparing Graft-first to Fistula-first Strategies in Older Patients With Incident End-stage Kidney Disease
Brief Title: Graft-first Versus Fistula-first in Older Patients With End-stage Kidney Disease
Acronym: GEMSSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00050577; R03AG060178-02 (NIH)
Record Dates: First submitted 2018-05-03; First posted 2018-06-04 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2020-05

CONDITIONS: Kidney Diseases
Keywords: graft; fistula; hemodialysis; Vascular access
MeSH Terms: conditions — Kidney Diseases; Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper extremity arteriovenous graft (AVG) - first (Experimental): Participants randomized to receive an AVG will undergo surgery to have an AVG placed.
  Interventions: Procedure: Upper arm arteriovenous graft surgery
- Upper extremity arteriovenous fistula (AVF) - first (Active Comparator): Participants randomized to receive an AVF will undergo surgery to have an AVF created.
  Interventions: Procedure: Upper arm arteriovenous fistula surgery

INTERVENTIONS:
Procedure: Upper arm arteriovenous graft surgery — Creation of arteriovenous graft vascular access for hemodialysis
  Arms: Upper extremity arteriovenous graft (AVG) - first
Procedure: Upper arm arteriovenous fistula surgery — Creation of arteriovenous fistula vascular access for hemodialysis
  Arms: Upper extremity arteriovenous fistula (AVF) - first

SUMMARY:
Many older adults require hemodialysis for advanced chronic kidney disease, but it is not clear which permanent vascular access method (fistula or graft) is best with respect to access effectiveness and patient satisfaction. In this pilot study, the study team will test the hypothesis that older adults undergoing graft access placement will more effectively transition from catheter-based to arteriovenous access-based hemodialysis; have fewer following vascular access procedures; have better upper extremity function; have better self-sufficiency with daily activities; and better health-related quality of life compared to those who undergo arteriovenous fistula access placement. The study will establish feasibility of randomizing older adults to the two types of arteriovenous access surgeries; evaluate relationships between measurements of pre-operative physical function and vascular access development; compare vascular access outcomes between the two groups; and gather longitudinal assessments of upper extremity muscle strength, performance of activities of daily living, and patients' reports of satisfaction with their vascular access and quality of life.

DETAILED DESCRIPTION:
Each year, more than 600,000 people in the United States receive life-saving hemodialysis (HD) treatments for end-stage kidney disease (ESKD), a third of whom are older adults.Timely placement of an arteriovenous (AV) vascular access (native AV fistula [AVF] or prosthetic AV graft [AVG]) is necessary to avoid (or limit) the use of tunneled central venous catheters (TCVC) for HD. 'Fistula First Catheter Last' national guidelines require placement of AVF as the AV access of first choice in all patients to achieve better patient survival. However, the benefits of AVF over AVG are least certain in older adults, as age-related biological changes independently modulate patient outcomes. Nationally representative cohort studies of older adults with incident ESKD have shown similar patient survival between those whose first AV access placed or used was a fistula or a graft.Compared with grafts, fistulas fail more often and necessitate longer times and more subsequent procedures to aid development, exposing older patients to time-consuming procedures that may negatively affect upper extremity strength and erode their quality of life. The contribution of pre-operative physical function to AV access outcomes and the impact of AV access placement on upper extremity strength and self-sufficiency have not been evaluated. This pilot trial will involve older adults with pre-dialysis advanced chronic kidney disease (CKD) or incident ESKD using a TCVC for HD who had no prior AV access surgery and have upper extremity vasculature suitable for either fistula or graft placement. Participants will be randomized to receive an upper extremity AVF-first or AVG-first access for HD. The primary objective of this pilot trial is to prospectively evaluate patient and vascular access outcomes in a randomized intervention and in a patient population in whom fistula-first guidelines have been applied despite the lack of proven benefit and at the detriment of more access failures and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* End-stage kidney disease (ESKD) on chronic hemodialysis (HD)
* Tunneled central venous catheter (TCVC) is the sole vascular access used for HD
* Advanced chronic kidney disease (CKD) expected to require HD initiation within 90 days of screening and deemed medically necessary by the treating nephrologist to proceed with arteriovenous (AV) access placement in preparation for HD initiation
* Did not undergo AV access placement in the past
* Medically eligible to receive AV fistula (AVF) or AV graft (AVG) placement as deemed by the treating nephrologist
* Surgically eligible to receive either an AVF or an AVG as deemed by the vascular surgeon
* HD is the intended long-term modality of treatment for ESKD
* Planning to remain within Wake Forest provided health care for at least 12 months

Exclusion Criteria:

* Presence of an AVF or AVG
* Previous attempt(s) for AV vascular access placement
* Native vasculature not suitable for placement of AV access
* Imminent transplant planned (within 6 months)
* Anticipated life expectancy <9 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Murea, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results obtained in the pilot trial, deidentified.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following the first article publication that stems from this pilot trial.
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of data has been approved by an independent review party identified for this purpose.

REFERENCES:
- [Background] Murea M, Burkart J. Finding the right hemodialysis vascular access in the elderly: a patient-centered approach. J Vasc Access. 2016 Sep 21;17(5):386-391. doi: 10.5301/jva.5000590. Epub 2016 Aug 1. PMID 27516143
- [Background] Yuo TH, Chaer RA, Dillavou ED, Leers SA, Makaroun MS. Patients started on hemodialysis with tunneled dialysis catheter have similar survival after arteriovenous fistula and arteriovenous graft creation. J Vasc Surg. 2015 Dec;62(6):1590-7.e2. doi: 10.1016/j.jvs.2015.07.076. Epub 2015 Sep 12. PMID 26372193
- [Background] Lok CE, Allon M, Moist L, Oliver MJ, Shah H, Zimmerman D. Risk equation determining unsuccessful cannulation events and failure to maturation in arteriovenous fistulas (REDUCE FTM I). J Am Soc Nephrol. 2006 Nov;17(11):3204-12. doi: 10.1681/ASN.2006030190. Epub 2006 Sep 20. PMID 16988062
- [Background] Peterson WJ, Barker J, Allon M. Disparities in fistula maturation persist despite preoperative vascular mapping. Clin J Am Soc Nephrol. 2008 Mar;3(2):437-41. doi: 10.2215/CJN.03480807. Epub 2008 Jan 30. PMID 18235150
- [Background] Woo K, Goldman DP, Romley JA. Early Failure of Dialysis Access among the Elderly in the Era of Fistula First. Clin J Am Soc Nephrol. 2015 Oct 7;10(10):1791-8. doi: 10.2215/CJN.09040914. Epub 2015 Aug 7. PMID 26254301
- [Background] Vascular Access 2006 Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S176-247. doi: 10.1053/j.ajkd.2006.04.029. No abstract available. PMID 16813989
- [Background] DeSilva RN, Patibandla BK, Vin Y, Narra A, Chawla V, Brown RS, Goldfarb-Rumyantzev AS. Fistula first is not always the best strategy for the elderly. J Am Soc Nephrol. 2013 Jul;24(8):1297-304. doi: 10.1681/ASN.2012060632. Epub 2013 Jun 27. PMID 23813216
- [Background] Richardson AI 2nd, Leake A, Schmieder GC, Biuckians A, Stokes GK, Panneton JM, Glickman MH. Should fistulas really be first in the elderly patient? J Vasc Access. 2009 Jul-Sep;10(3):199-202. doi: 10.1177/112972980901000311. PMID 19670174
- [Derived] Robinson T, Geary RL, Davis RP, Hurie JB, Williams TK, Velazquez-Ramirez G, Moossavi S, Chen H, Murea M. Arteriovenous Fistula Versus Graft Access Strategy in Older Adults Receiving Hemodialysis: A Pilot Randomized Trial. Kidney Med. 2021 Feb 10;3(2):248-256.e1. doi: 10.1016/j.xkme.2020.11.016. eCollection 2021 Mar-Apr. PMID 33851120
- [Derived] Murea M, Geary RL, Houston DK, Edwards MS, Robinson TW, Davis RP, Hurie JB, Williams TK, Velazquez-Ramirez G, Bagwell B, Tuttle AB, Moossavi S, Rocco MV, Freedman BI, Williamson JD, Chen H, Divers J. A randomized pilot study to evaluate graft versus fistula vascular access strategy in older patients with advanced kidney disease: results of a feasibility study. Pilot Feasibility Stud. 2020 Jun 17;6:86. doi: 10.1186/s40814-020-00619-9. eCollection 2020. PMID 32551134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Started | 23 | 21
Completed | 18 | 21
Not Completed | 5 | 0
Not completed — Surgery Cancelled | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Received different surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Full Range); unit: years] | 72.8 [71.1 to 82.0] | 78.9 [70.7 to 81.1] | 76.3 [70.8 to 81.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 12 | 15 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility- Eligibility for Randomization
Description: Proportion of screened participants deemed eligible for randomization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Group: Group includes all Participants that signed Consent
Arm/Group | Total Group
Number analyzed (Participants) | 77
Participants | 54

2. Primary Outcome: Feasibility- Consent to Randomization
Description: Proportion of eligible participants who consent to randomization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Group Randomized: All Participants that signed Consent to Randomization
Arm/Group | Total Group Randomized
Number analyzed (Participants) | 54
Participants | 44

3. Primary Outcome: Feasibility- AV Graft or Fistula Placement
Description: Proportion of participants who undergo AV graft or fistula placement within 90 days of randomization.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 23 | 21
Participants | 18 | 21

4. Secondary Outcome: Upper Extremity Strength
Description: The grip-strength test will be performed twice on each hand for each assessment and the mean of the two results will be used for statistical analyses; a cut-off point <16 kg in women and <26 kg in men will define muscle weakness. Changes in grip strength will be compared between the two access interventions. Assessed with upper arm grip-strength test in each arm using a hand-held dynamometer.
Time Frame: 3 and 6 months
Population: Subject could not move hand from past stroke; Subject had joint pain; not completed due to distance
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
kilograms
  3 Months | 21.3 (5.6) | 22.6 (6.4)
  6 Months: number analyzed (Participants) | 11 | 12
  6 Months | 19.1 (6.7) | 20.4 (7.2)
  Baseline | 19.6 (3.3) | 17.4 (3.5)

5. Secondary Outcome: Patient Satisfaction With Vascular Access
Description: Vascular access questionnaire will be used to assess differences in patient satisfaction with vascular access between the two access interventions using the short-form vascular access questionnaire (SF-VAQ). Mean scores obtained on SF-VAQ will be compared. SF-VAQ score range 4 -20 with higher scores indicating more satisfaction with the vascular access.
Time Frame: 3 and 6 months
Population: Number differ form total number of randomized, 1 participant expired, not all questionnaires collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 16 | 19
score on a scale
  3 months: number analyzed (Participants) | 8 | 19
  3 months | 9.75 (3.45) | 8.82 (1.53)
  6 Months: number analyzed (Participants) | 16 | 8
  6 Months | 7.55 (2.74) | 8.75 (1.16)
  week 2 | 10.1 (3.18) | 9.21 (2.39)

6. Secondary Outcome: Performance on Activities of Daily Living (ADLs)
Description: The level of independence will be evaluated using ADLs. ADL score range 0-30, with higher scores denoting more dependence on other people to perform the usual daily activities.
Time Frame: Baseline and 6 months
Population: Patients declined survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 4.5 (1.6) | 4.75 (1.28)
  Month 6: number analyzed (Participants) | 8 | 8
  Month 6 | 4.2 (1.82) | 5.11 (1.16)

7. Secondary Outcome: Performance on Activities of Instrumental Daily Living ADLs (IADLs)
Description: The level of independence will be evaluated using IADLs instruments. ADL score range 0-31, with higher scores denoting more dependence on other people.
Time Frame: Baseline, 3 and 6 months
Population: Patients declined survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 14 | 17
score on a scale
  Baseline | 5.28 (2.49) | 4.5 (1.45)
  Month 6: number analyzed (Participants) | 9 | 7
  Month 6 | 4.4 (2.65) | 6.42 (2.64)

8. Secondary Outcome: Depression
Description: Depression scores assessed with the patient health questionnaire (PHQ-9) will be compared between the two vascular access arms. PHQ-9 score range 0-27. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Time Frame: 3 and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Health-related Quality of Life (HRQoL) - Mental Health (MCS-12) Scores
Description: The impact of the two types of vascular access on HRQoL will be assessed using the Kidney Disease Quality of Life Short Form (KDQOL-SF) version 1.3. which consists of a generic core (Short Form-36 [SF-36]) and an 11-item kidney disease-specific scale. Score range 0 to 100, with higher scores reflecting better quality of life.
Time Frame: Baseline, Month 3, and Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 15 | 19
score on a scale
  Month 3 | 54.38 (13.26) | 46.27 (5.66)
  Month 6 | 53.79 (17.31) | 58.2 (5.91)
  Baseline | 53.38 (8.05) | 51.46 (11.37)

10. Secondary Outcome: Health-related Quality of Life (HRQoL) - Physical Health (PCS-12) Scores
Description: as for outcome 9
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 15 | 19
score on a scale
  Month 3 | 39.02 (8.45) | 39.44 (5.23)
  Month 6 | 40.77 (7.73) | 36.12 (5.55)
  Baseline | 29.89 (12.09) | 36.75 (10.7)

11. Secondary Outcome: Physical Activity Level
Description: The Rapid Assessment of Physical Activity (RAPA) instrument will be used to assess habitual physical activity. RAPA test score ≤ 3 corresponded to a sedentary lifestyle or a very light activity level; values ≥4 indicated a moderate to vigorous active lifestyle.
Time Frame: 3 and 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Physical Activity Level 4-meter Gait
Description: The 4MGS test is a simple screening test and a useful predictor of worsening daily activity in patients with chronic respiratory diseases.
Time Frame: Baseline, month 3 and 6
Population: Assessment was added on 2.4.2019 - Subjects could not walk un-assisted
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 5 | 10
meters per second
  Baseline: number analyzed (Participants) | 3 | 10
  Baseline | 7.5 (3.04) | 5.1 (1.61)
  Month 3: number analyzed (Participants) | 5 | 7
  Month 3 | 6.88 (2.23) | 6.04 (2.36)
  Month 6: number analyzed (Participants) | 5 | 7
  Month 6 | 5.74 (1.15) | 6.34 (2.45)

13. Secondary Outcome: Number of Subjects With No Pain at the AV Access Site
Description: This will be determined by using the Verbal Descriptor Scale (VDS). The Verbal Descriptor Scale (VDS) is comprised of a series of descriptive phrases that refer to different levels of pain severity or intensity. Patients select the phrase that best describes their current pain - The verbal descriptor scale asks the patient to describe her or his pain using the following descriptors: "no pain," "mild pain," "moderate pain," "severe pain," or "pain as bad as it could be."
Time Frame: Baseline, 3 and 6 months
Population: Patient expired, some participants also declined (at times) answering questions, and some visits were not performed due to travel distance
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 17 | 19
Participants
  Baseline | 6 | 13
  Month 3: number analyzed (Participants) | 8 | 11
  Month 3 | 4 | 10
  Month 6: number analyzed (Participants) | 9 | 8
  Month 6 | 7 | 7

14. Secondary Outcome: Number of Subjects With Mild Pain at the AV Access Site
Description: as for outcome 13
Time Frame: Baseline, Month 3 and Month 6
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 17 | 19
Participants
  Baseline | 6 | 1
  Month 3: number analyzed (Participants) | 8 | 11
  Month 3 | 2 | 1
  Month 6: number analyzed (Participants) | 9 | 8
  Month 6 | 0 | 0

15. Secondary Outcome: Number of Subject With Moderate Pain at the AV Access Site
Description: as for outcome 13
Time Frame: Baseline, Month 3 and Month 6
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 17 | 19
Participants
  Baseline | 3 | 5
  Month 3: number analyzed (Participants) | 8 | 11
  Month 3 | 2 | 0
  Month 6: number analyzed (Participants) | 9 | 8
  Month 6 | 2 | 1

16. Secondary Outcome: Number of Subjects With Severe Pain at the AV Access Site
Description: as for outcome 13
Time Frame: Baseline, Month 3 and Month 6
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 17 | 19
Participants
  Baseline | 2 | 0
  Month 3: number analyzed (Participants) | 8 | 11
  Month 3 | 0 | 0
  Month 6: number analyzed (Participants) | 9 | 8
  Month 6 | 0 | 1

17. Other Pre Specified Outcome: AV Access Primary Failure
Description: Rate of AV access primary failure between the two AV access strategies. Primary access failure is defined as permanent failure of the fistula or graft before hemodialysis suitability. This will include inadequate maturation, thrombosis, failure of first and subsequent cannulations, and/or other complications leading to nonfunctional fistula or graft.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
Participants | 4 | 5

18. Other Pre Specified Outcome: AV Access Infection
Description: Incidence rate of AV access infection between the two AV access strategies. This will include fistula or graft cellulitis, abscess, and/or bacteremia due to AV access infection.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
Participants | 3 | 2

19. Other Pre Specified Outcome: AV Access Successful Cannulation
Description: Will compare the proportion of patients with successful AV access cannulation between the two AV access strategies. Successful cannulation is defined by the use of the AV access as the primary vascular access for hemodialysis (the fistula or graft access has been cannulated with two 16- or 15-gauge needles for ≥3 consecutive dialysis sessions and the dialysis central venous catheter was removed).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
Participants | 8 | 8

20. Other Pre Specified Outcome: AV Access Secondary Failure
Description: Rate of AV access secondary failure between the two AV access strategies. Secondary access failure is defined by permanent AV access failure after the fistula or graft met dialysis suitability criteria with subsequent abandonment.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 18 | 21
Participants | 5 | 8

21. Other Pre Specified Outcome: AV Access Procedures - Number of Surgical Re-intervention on Index AV Access Procedures
Description: Number of AV access procedures per 100 patient-days between the two AV access strategies. This will include angioplasty, thrombectomy, stent placement, repeat surgery, and/or surgical superficialization.
Time Frame: 12 months
Measure: Number; unit: procedures per 100 patient-days
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
procedures per 100 patient-days | 3 | 4

22. Other Pre Specified Outcome: AV Access Procedures - Number of Endovascular Interventions on Index AV Procedures Access
Description: as for outcome 21
Time Frame: 12 months
Measure: Number; unit: procedures per 100 patient-days
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
Number analyzed (Participants) | 13 | 16
procedures per 100 patient-days | 5 | 7

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Upper Extremity Arteriovenous Graft (AVG) - First | Upper Extremity Arteriovenous Fistula (AVF) - First
All-Cause Mortality (participants affected / at risk) | 3/23 | 2/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 1/23 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upper Extremity Arteriovenous Graft (AVG) - First (N=23) | Upper Extremity Arteriovenous Fistula (AVF) - First (N=21)
catheter-related infection (Infections and infestations) | 1 (1) | 0 (0) — one had a catheter-related infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03545113/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03545113/ICF_002.pdf